CLINICAL TRIAL: NCT05136144
Title: Open-Label Adaptive Design Study to Explore the Safety and Efficacy of Multiple Treatment Regimens With the Akt Inhibitor SM-020 Gel in 1.0% and 0.1% Gel Formulations in Subjects With Seborrheic Keratosis
Brief Title: Adaptive Design Study for Safety and Efficacy of Treatment Regimens With SM-020 in Subjects With Seborrheic Keratosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: DermBiont, Inc. (Industry)
Collaborators: Zepeda Dermatologia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DBI-SM-201
Record Dates: First submitted 2021-11-08; First posted 2021-11-29 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Seborrheic Keratosis
MeSH Terms: conditions — Keratosis, Seborrheic

STUDY DESIGN:
Intervention Model Description: Adaptive design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SM-020 (Experimental): Topical Akt Inhibitor SM-020 Gel
  Interventions: Drug: SM-020

INTERVENTIONS:
Drug: SM-020 — Topical Akt Inhibitor SM-020 Gel

SUMMARY:
This is a first-in-humans adaptive design open label trial to explore the safety and efficacy of SM-020. Multiple dosing cohorts will be enrolled. The first cohort will have a two-week treatment period of twice daily applications followed by a four-week follow-up period. Based on the results at any time from the first and subsequent cohorts, additional cohorts will explore different dosing regimens.

DETAILED DESCRIPTION:
This is a first-in-humans adaptive design open label trial to explore the safety and efficacy of SM-020. Multiple dosing cohorts will be enrolled. The first cohort will have a two-week treatment period of twice daily applications followed by a four-week follow-up period. Based on the results at any time from the first and subsequent cohorts, additional cohorts will explore different dosing regimens.

Variables to be considered in the design of cohorts include frequency of application and duration of application.

The maximum duration of a treatment period is 12 weeks for any subject.

35 Subjects have been enrolled to date in the following 7 cohorts:

Cohort 1: SM-020 gel 1.0% BID (Bis in die) for 14 days

Cohort 2: SM-020 gel 1.0% BID for 28 days

Cohort 3: SM-020 gel 1.0% BID pulsed dosing 4 days on/4 days off

Cohort 4: SM-020 gel 1.0% BID for 28 days to facial SKs

Cohort 5: SM-020 gel 1.0% TIW (Three times a week) under occlusion for 28 days

Cohort 6: SM-020 gel 1.0% BID for 28 days with intertriginous SKs

Cohort 7: SM-020 gel 0.1% BID for 28 days to facial SKs

Anticipated subsequent cohorts to be enrolled:

Cohort 8: SM-020 gel 1.0% BID for 56 days

Cohort 9: SM-020 gel 1.0% BID for 28 days

Cohort 10: SM-020 gel 1.0% QD (Quaque die) for 28 days

Cohort 11: SM-020 gel 0.1% BID for 28 days

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to comprehend and willing to sign an informed consent form (ICF).
2. At least 18 years of age.
3. Must have a minimum of 5 eligible facial, truncal, intertriginous, or extremity SKTLs. A maximum of 10 will be targeted for treatment. There will be a maximum of 5 PLA 2's per subject. An eligible SKTL must each:

   1. Have one or more of the following clinical features throughout the entirety of the lesion consistent with SKs: stuck-on, warty, waxy, scaly, milia-like cyst, tan to black
   2. For subjects randomized for assessment with clinical diagnosis and dermoscopy, SKs must also have one or more of the dermoscopy features throughout the entirety of the lesion: moth-eaten border, fingerprinting structures, network-like pattern, network pattern, crypts (comedo-like openings), milia cysts, pinpoint vessels, hairpin vessels, fat fingers, sharp demarcation, blue-white pigmentation, more than one color, cerebriform structure, irregular, polymorphic pattern, fissures, white artefacts, irregular vessels (Simionescu et al., 2012).
   3. Have a Physician's Lesion Assessment (PLA) of 2 (a thickness that is ≤1mm) or 3 (a thickness that is >1mm)
   4. Have a greatest diameter that is ≥5mm and ≤15mm
   5. Be a discrete, well-defined, separate lesion
   6. Not be covered with hair which, in the Investigator's opinion, would interfere with the study gel treatment or the study evaluations
   7. Not be pedunculated
   8. Not be on the eyelid
   9. Not be within 5mm of the orbital rim
4. Must be free of any known disease state or physical condition which, in the Investigator's opinion, might impair evaluation of any SKTL or which exposes the subject to an unacceptable risk by study participation.
5. Must be willing and able to follow all study instructions and to attend all study visits.
6. As applicable, technical ability and willingness to apply Investigational Product (IP).
7. Must be willing to have all partial, incompletely, or non-responding SKTLs removed surgically by shave excision during the final visit.

Exclusion Criteria:

1. Positive urine pregnancy test, pregnant, lactating, or female of childbearing potential who does not agree to use an active method of birth control for the duration of the study.
2. SK lesions that are clinically atypical and/or rapidly growing in size.
3. Presence of multiple eruptive SK lesions (sign of Leser-Trelat).
4. Current systemic malignancy.
5. Any use of the following systemic therapies within the specified period, or unwilling to meet the following washouts, prior to the Baseline visit:

   1. Retinoids; 180 days
   2. Glucocorticosteroids; 28 days
   3. Anti-metabolites (e.g., methotrexate); 28 days
6. Any use of the following topical therapies within the specified period, or unwilling to meet the following washouts, prior to the Baseline visit and while on study on, or in a proximity to any SKTL that, in the Investigator's opinion, could interfere with the investigational product study treatment applications or the study assessments:

   1. Laser, light or other energy-based therapy [e.g., intense pulsed light (IPL), photo-dynamic therapy (PDT)]; 180 days
   2. Liquid nitrogen, electrodesiccation, curettage, imiquimod, 5-fluorouracil, or ingenol mebutate; 60 days
   3. Retinoids; 28 days
   4. Microdermabrasion or superficial chemical peels; 14 days
   5. Glucocorticosteroids or antibiotics; 14 days
7. Occurrence or presence of any of the following within the specified period prior to the Baseline visit on or in the proximity of any SKTL that, in the Investigator's opinion, could interfere with the investigational product study treatment applications or the study assessments:

   1. Cutaneous malignancy; 180 days
   2. Sunburn; currently
   3. A pre-malignancy (e.g., actinic keratosis); currently
   4. Body art (e.g., tattoos, piercing, etc.); currently
8. History of sensitivity to any of the ingredients in the investigational product.
9. Any current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage, etc.), or other condition(s) (e.g., sunburn, excessive hair, open wounds, lupus, photosensitive disorders etc.) that, in the opinion of the Investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations.
10. Participation in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to the Screening visit.
11. History of hypertrophic scarring or keloid formation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Superiority of 56-day BID treatment with SM-020 gel 1.0% over 28-day BID treatment with SM-020 gel 1.0% | Through 20 weeks
  Measured by the proportion of all SKTLs (Seborrheic Keratosis Target Lesion) that achieve clearance (PLA score of 0) at final study visit
Superiority of 28-day BID treatment with SM-020 gel 1.0% over 28-day QD treatment with SM-020 gel 1.0% | Through 20 weeks
  Measured by the proportion of all SKTLs that achieve clearance (PLA score of 0)
Superiority of 28-day BID treatment with SM-020 gel 1.0% over 28-day BID treatment with SM-020 gel 0.1% | Through 20 weeks
  Measured by the proportion of all SKTLs that achieve clearance (PLA score of 0)

SECONDARY OUTCOMES:
Superiority of 56-day BID treatment with SM-020 gel 1.0% over 28-day BID treatment with SM-020 gel 1.0% | Through 20 weeks
  Measured by the proportion of facial SKTLs, truncal SKTLs, intertriginous SKTLs, and extremity SKTLs that achieve clearance (PLA score of 0)
Superiority of 56-day BID treatment with SM-020 gel 1.0% over 28-day BID treatment with SM-020 gel 1.0% | Through 20 weeks
  Measured by the proportion of all SKTLs, facial SKTLs, truncal SKTLs, intertriginous SKTLs, and extremity SKTLs with a PLA of 0 or 1
Superiority of 56-day BID treatment with SM-020 gel 1.0% over 28-day BID treatment with SM-020 gel 1.0% | Through 20 weeks
  Measured by the proportion of subjects achieving clearance of all SKTLs, facial SKTLs, truncal SKTLs, intertriginous SKTLs, and extremity SKTLs
Superiority of 56-day BID treatment with SM-020 gel 1.0% over 28-day BID treatment with SM-020 gel 1.0% | Through 20 weeks
  Measured by the proportion of subjects achieving clearance of at least 5 of all SKTLs
Superiority of 56-day BID treatment with SM-020 gel 1.0% over 28-day BID treatment with SM-020 gel 1.0% | Through 20 weeks
  Measured by the proportion of all SKTLs/subject, facial SKTLs/subject, truncal SKTLs/subject, intertriginous SKTLs/subject, and extremity SKTLs/subject achieving a PLA of 0
Superiority of 56-day BID treatment with SM-020 gel 1.0% over 28-day BID treatment with SM-020 gel 1.0% | Through 20 weeks
  Measured by the proportion of all SKTLs, facial SKTLs, truncal SKTLs, intertriginous SKTLs, and extremity SKTLs with a SSA (Subject's Self-Assessment) of 0 or 1
Superiority of 56-day BID treatment with SM-020 gel 1.0% over 28-day BID treatment with SM-020 gel 1.0% | Through 20 weeks
  Measured by the proportion of all SKTLs, facial SKTLs, truncal SKTLs, intertriginous SKTLs, and extremity SKTLs with a SSA of 0
Superiority of 56-day BID treatment with SM-020 gel 1.0% over 28-day BID treatment with SM-020 gel 1.0% | Through 20 weeks
  Measured by the percent recurrence of all SKTLs, facial SKTLs, truncal SKTLs, intertriginous SKTLs, and extremity SKTLs

CONTACTS AND LOCATIONS:
Overall Officials: David Zepeda, MD, Principal Investigator — Zepeda Dermatologia
Locations (1):
- Zepeda Dermatologia, Santa Tecla, La Libertad Department, El Salvador

IPD SHARING:
Plan to Share IPD: No